CLINICAL TRIAL: NCT07262853
Title: Examining the Effectiveness of a Dual Executive Function Training Package: Protocol for a Randomised Controlled Trial
Brief Title: Dual Executive Function Training Package
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The Good Shepherd Project
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: ADHD; Dyslexia; Autism
Keywords: Executive Functions; intervention; attention-deficit/hyperactivity disorder; specific learning difficulties; autism spectrum disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dyslexia; Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial will be adopted in which all assessors are blinded to the treatment condition of the students. Participants will be randomly assigned to either an experimental or a waitlist control group, stratified by diagnosis. Each intervention group (n = 48) will receive the dual EF training programme, while corresponding waitlist controls (n = 48) will receive it after the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental: ADHD Group (Experimental): This experimental group will receive the executive function training in primary schools in Hong Kong.
  Interventions: Other: Executive Function Training
- Experimental: RD Group (Experimental): This experimental group will receive the executive function training in primary schools in Hong Kong.
  Interventions: Other: Executive Function Training
- Experimental: ASD Group (Experimental): This experimental group will receive the executive function training in primary schools in Hong Kong.
  Interventions: Other: Executive Function Training
- Waitlist Control: ADHD Group (No Intervention): Students assigned to the waitlist control group will receive the executive function training program after the experimental group has completed it.
- Waitlist Control: RD Group (No Intervention): Students assigned to the waitlist control group will receive the executive function training program after the experimental group has completed it.
- Waitlist Control: ASD Group (No Intervention): Students assigned to the waitlist control group will receive the executive function training program after the experimental group has completed it.

INTERVENTIONS:
Other: Executive Function Training — All students will participate in a structured EF training program designed to support those with SENs. The EF training program will include weekly group training sessions lasting one hour each, which will be organised in small groups of six students to foster interaction and peer support.
  Arms: Experimental: ADHD Group; Experimental: ASD Group; Experimental: RD Group

SUMMARY:
Executive function (EF) refers to the cognitive processes that enable goal-directed regulation of thoughts, emotions, and behaviours. Two interrelated domains are commonly distinguished: "cool" EF, which involves abstract cognitive processes, and "hot" EF, which involves regulation in emotionally or motivationally charged contexts. Children with special educational needs (SENs) frequently show difficulties across both domains, yet most interventions target one in isolation. The present study aims to evaluate the effectiveness of a dual EF training package for three of the most prevalent SENs groups: attention-deficit/hyperactivity disorder (ADHD), specific learning difficulties (SpLD), and autism spectrum disorder (ASD). A total of 288 primary school students aged 6-12 years with a diagnosis of ADHD, ASD, or SpLD will be recruited. Participants will be randomly assigned to either an intervention or waitlist control group, stratified by diagnosis. Each intervention group (n = 48) will receive the dual EF training programme, while corresponding waitlist controls (n = 48) will receive it after the study. Pre- and post-intervention assessments will include neuropsychological tests of EF, teacher- and parent-reported behavioural ratings, and measures of disability impact, school satisfaction, and social participation.

DETAILED DESCRIPTION:
Executive functions (EF) are a set of higher-order cognitive processes that enable children to regulate their thoughts, emotions, and behaviours in pursuit of goals. Core domains include working memory, inhibitory control, and cognitive flexibility, often referred to as cool EF because they are typically measured in abstract, decontextualised contexts. Cold EFs are top-down cognitive processes that are logically based or mechanistic and operate in affectively neutral contexts. In contrast, hot EF refers to regulation in affectively or motivationally charged situations, encompassing delay discounting, affective/risky decision-making, and interpersonal and social behaviour. Both domains are crucial for children's learning, adaptation, and participation, but they rely on partially distinct neural systems and show different developmental trajectories. Importantly, recent models emphasise that hot and cool EF should not be viewed as isolated constructs but rather as interconnected components along a continuum. In real-world learning and social contexts, cognitive and affective demands are often intertwined. For example, sustaining working memory while managing frustration, or planning actions while negotiating peer dynamics, highlighting the need for interventions that address both hot and cool domains simultaneously.

EF difficulties are particularly salient in the context of special educational needs (SENs). Children with SENs are disproportionately likely to present with impairments in both hot and cool EF, which underpin many of the learning and behavioural challenges they face in schools. Among these, attention-deficit/hyperactivity disorder (ADHD), autism spectrum disorder (ASD), and specific learning difficulties (SpLD) are the three most prevalent conditions worldwide, and they are consistently associated with executive dysfunction. ADHD, ASD, and SpLD are all characterised by combined hot and cool EF deficits. In ADHD, cool EF weaknesses in working memory, inhibition, and sustained attention are compounded by hot EF problems such as poor delay of gratification, impulsivity, and emotional dysregulation. ASD presents with cool EF impairments in flexibility, planning, and working memory. It also shows hot EF deficits in emotional regulation, reward processing, and theory of mind. SpLD is often framed as academic skill deficits. However, it also involves cool EF challenges in working memory, processing speed, and attention as well as hot EF challenges related to frustration tolerance and motivation. Despite this dual profile, many existing interventions have focused disproportionately on one side of the EF spectrum, typically emphasising cool EF while neglecting hot EF. To provide meaningful support for children with SENs, a more comprehensive approach is needed, one that systematically integrates both domains.

Existing EF interventions provide partial solutions but leave important gaps. Cognitive training studies, such as Re et al. (2015) have demonstrated that children with ADHD symptoms can improve in attention, inhibition, and working memory following structured training. These domains reflect cool EF, and while the programme successfully enhanced cognitive performance, the gains were largely confined to laboratory tasks, with modest evidence of generalisation to socio-emotional or classroom functioning. Hot EF, such as emotional regulation or social reasoning, was not directly addressed. A more ecological approach is seen in the Cognitive-Functional (Cog-Fun) intervention for ADHD. Cog-Fun is an occupational therapy programme that emphasises metacognitive strategy use, planning, organisation, and self-monitoring in daily life. Parents are also coached to support the application of strategies at home. While Cog-Fun is effective in improving organisation, homework performance, and children's self-directed behaviour, its focus remains on cool EF, with only indirect influence on hot EF domains such as emotional regulation and motivation through parent involvement.

More recent work has explicitly attempted to integrate hot EF. Shuai et al. (2017) developed an EF training package for children with ADHD that included not only core cool EF skills (working memory, inhibition, planning, flexibility, and verbal fluency) but also hot EF components such as emotional regulation. Their results showed improvements in both cognitive control and social understanding, underscoring the value of a dual-domain approach. However, the scope of hot EF was narrow, confined to Theory of Mind tasks and behavioural ratings of emotional control, and the programme was delivered in a clinic-based format, limiting scalability and ecological validity in school contexts. Similarly, Jasni et al. (2025) implemented a psychosocial group intervention combining cognitive skills training with social skills and emotional regulation exercises. Although not framed explicitly in hot-cool EF terms, the programme recognised the importance of targeting both domains. Children showed improvements in EF performance and social behaviour. Yet, the hot EF elements were integrated only loosely with cognitive training, and the lack of a systematic framework to connect the two domains limited the intervention's conceptual clarity and generalisability.

Research on EF interventions in ASD and specific learning disabilities (SpLD) reveals similar limitations. For ASD, interventions often focus on improving planning, flexibility, and organisation through structured tasks or cognitive-behavioural strategies, targeting cool EF deficits. Some studies incorporate social skills training, which overlaps with hot EF, but these are typically run as separate programmes rather than integrated EF training. This fragmented approach fails to address the interdependence of cognitive and socio-emotional regulation, both of which are impaired in ASD. In SpLD, interventions predominantly target working memory, inhibition, or attention to support reading or mathematics performance. These cool EF-focused programmes have demonstrated efficacy in improving task-related outcomes, but they neglect hot EF processes such as self-regulation, frustration tolerance, and motivational control, which are equally important for sustaining learning in students with SpLD. The absence of a hot EF component leaves a gap in addressing the broader challenges faced by students with SpLD in daily classroom participation.

Together, these findings demonstrate that while ADHD, ASD, and SpLD are all characterised by combined deficits in hot and cool EF, most existing interventions are narrow in scope, either focusing almost exclusively on cool EF or including only partial and unsystematic coverage of hot EF. Furthermore, interventions are often delivered in clinical rather than classroom contexts, which constrains ecological validity and limits opportunities for students to practise EF in authentic academic and social environments. These limitations highlight the need for a comprehensive, classroom-based intervention that systematically integrates both hot and cool EF domains, such as the Dual EF Training Package described in the present study.

Existing EF interventions have tended to adopt a fragmented architecture, with cool and hot EF components treated as separate strands rather than as interdependent processes. Cognitive training programmes often prioritise laboratory-based tasks of working memory, inhibition, or flexibility, while socio-emotional curricula focus on behavioural regulation or social skills, but the two are rarely integrated within a coherent structure. This separation is at odds with contemporary models conceptualising EF as a continuum, where cognitive and affective regulation are dynamically interlinked. In everyday contexts, children must simultaneously hold information in mind, resist distraction, and adapt flexibly, while also regulating frustration, negotiating peer relationships, and maintaining motivation. An intervention that addresses only one side of this continuum risks producing narrow, domain-bound effects with limited generalisation.

Theoretical and empirical precedents suggest that integration is both necessary and feasible. Frameworks such as the expected value of control model highlight how motivational and affective signals shape the allocation of cognitive control, underscoring the need to co-train these systems under one united topic. Similarly, approaches in self-regulated learning and early childhood curricula such as Tools of the Mind demonstrate the benefits of coupling cognitive strategies with emotion regulation and motivational scaffolding under the same area of focus. Yet, most existing efforts remain partial, addressing affect only indirectly or situating cognitive and affective training in parallel modules rather than within a unified sequence.

Taken together, prior studies demonstrate that EF is malleable and that both cognitive and socio-emotional interventions can yield measurable benefits. However, they also reveal persistent limitations: most interventions either focus narrowly on cool EF or address hot EF only incidentally, and few are implemented in ecologically valid, classroom-based contexts. The current study seeks to evaluate the effectiveness of a dual EF Training Package designed to address these gaps by explicitly integrating cool and hot EF within a coherent, school-based curriculum. The programme adopts a theme-based, paired structure in which each cool EF skill is systematically linked to its hot EF counterpart within the same chapter. To our knowledge, it represents the first intervention to employ a systematically matched hot-cool EF design across an entire curriculum. This theoretically grounded and ecologically valid model is expected to yield improvements not only in core EF performance but also in broader functional outcomes most relevant to children with SENs.

ELIGIBILITY:
Inclusion Criteria:

* aged between 6 and 11 years
* studying at primary schools in HK
* confirmed or suspected ADHD, ASD, or SpLD

Exclusion Criteria:

* received executive function training
* comorbid conditions

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 288 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Verbal Working Memory | One week before the intervention
  Verbal working memory will be assessed using the backward digit spans subtest from the third edition of the Wechsler Intelligence Scale for Children-Third Edition (WISC-III).
Verbal Working Memory | One week after the intervention
  Verbal working memory will be assessed using the backward digit spans subtest from the third edition of the Wechsler Intelligence Scale for Children-Third Edition (WISC-III).
Inhibition | One week before the intervention
  The Stroop color and word test is a widely used assessment for measuring inhibition. In this test, participants will be presented with colour words printed in mismatched ink colors (for example, the word "red" written in blue ink). They will be instructed to quickly name the ink colour of each word while ignoring the word's meaning. This effort to suppress the meaning of the word to identify the ink colour consistently leads to longer response times compared to naming the colour of congruent stimuli (such as "red" printed in red ink).
Inhibition | One week after the intervention
  The Stroop color and word test is a widely used assessment for measuring inhibition. In this test, participants will be presented with colour words printed in mismatched ink colors (for example, the word "red" written in blue ink). They will be instructed to quickly name the ink colour of each word while ignoring the word's meaning. This effort to suppress the meaning of the word to identify the ink colour consistently leads to longer response times compared to naming the colour of congruent stimuli (such as "red" printed in red ink).
Attentional Control and Cognitive Flexibility | One week before the intervention
  The contingency naming test will assess attentional control and cognitive flexibility through four rules of increasing difficulty, using a stimulus set that includes nine practice items and 27 test items. Each stimulus will consist of an outer shape (circle, triangle, or square) in various colors (blue, yellow, or red), along with a smaller independent shape (circle, triangle, or square) inside the outer shape. Some stimuli will feature a backward arrow positioned directly above the outer shape. Participants will be instructed to name the stimuli based on the rule level within a set time limit.
Attentional Control and Cognitive Flexibility | One week after the intervention
  The contingency naming test will assess attentional control and cognitive flexibility through four rules of increasing difficulty, using a stimulus set that includes nine practice items and 27 test items. Each stimulus will consist of an outer shape (circle, triangle, or square) in various colors (blue, yellow, or red), along with a smaller independent shape (circle, triangle, or square) inside the outer shape. Some stimuli will feature a backward arrow positioned directly above the outer shape. Participants will be instructed to name the stimuli based on the rule level within a set time limit.
School Satisfaction | One week before the intervention
  School satisfaction will be assessed using six items derived from the Longitudinal Study of Australian Children. Respondents will rate each item on a four-point Likert scale ranging from strongly agree to strongly disagree.
School Satisfaction | One week after the intervention
  School satisfaction will be assessed using six items derived from the Longitudinal Study of Australian Children. Respondents will rate each item on a four-point Likert scale ranging from strongly agree to strongly disagree.
Executive Function | One week before the intervention
  A short form of the Behavior Rating Inventory of Executive Function (BRIEF) includes questionnaires for both parents and teachers aimed at evaluating EF in home and school settings. The BRIEF contains 24 items, which produce eight scales: Initiate, working memory, plan/organise, organisation of materials, monitor, inhibit, shift, and emotional control. Parents and teachers will rate their child or student's behaviour on a 3-point Likert scale, ranging from 1 (never) to 3 (often).
Executive Function | One week after the intervention
  A short form of the Behavior Rating Inventory of Executive Function (BRIEF) includes questionnaires for both parents and teachers aimed at evaluating EF in home and school settings. The BRIEF contains 24 items, which produce eight scales: Initiate, working memory, plan/organise, organisation of materials, monitor, inhibit, shift, and emotional control. Parents and teachers will rate their child or student's behaviour on a 3-point Likert scale, ranging from 1 (never) to 3 (often).
Social Participation | One week before the intervention
  The Social Participation Questionnaire consists of 24 statements distributed across four subscales: Friendships/relationships (five items), contacts/interactions (nine items), student's social self-perception (five items), and acceptance by classmates (five items). Class teachers will complete the SPQ for the students by responding to the statements on a 5-point Likert-type scale, with options ranging from 1 (this does not apply at all) to 5 (this strongly applies).
Social Participation | One week after the intervention
  The Social Participation Questionnaire consists of 24 statements distributed across four subscales: Friendships/relationships (five items), contacts/interactions (nine items), student's social self-perception (five items), and acceptance by classmates (five items). Class teachers will complete the SPQ for the students by responding to the statements on a 5-point Likert-type scale, with options ranging from 1 (this does not apply at all) to 5 (this strongly applies).
Severity of Disability | One week before the intervention
  The severity of disability will be measured based on the seven domains of life: material well-being, health, safety, productive activity, place in community, intimacy, and emotional well-being. The seven items will be rated on a 5-point Likert scale, ranging from 1 (not at all affected) to 5 (extremely affected).
Severity of Disability | One week after the intervention
  The severity of disability will be measured based on the seven domains of life: material well-being, health, safety, productive activity, place in community, intimacy, and emotional well-being. The seven items will be rated on a 5-point Likert scale, ranging from 1 (not at all affected) to 5 (extremely affected).

CONTACTS AND LOCATIONS:
Locations (1):
- EdUHK, Tai Po, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share IPD is not yet finalized due to ethical consideration.